CLINICAL TRIAL: NCT01739361
Title: Phase IIa Randomized Controlled Trial of Acetaminophen for the Reduction of Oxidative Stress in Severe Sepsis
Brief Title: Acetaminophen for the Reduction of Oxidative Injury in Severe Sepsis
Acronym: ACROSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Janz, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APAP-121486
Record Dates: First submitted 2012-11-26; First posted 2012-12-03 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen (Experimental): Patients will receive acetaminophen at the dose of 1 gram by mouth or by enteral feeding tube every six hours for a total of 72 hours.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Patients will receive placebo by mouth or by enteral feeding tube every six hours for 72 hours.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acetaminophen
  Arms: Acetaminophen
Drug: placebo
  Arms: Placebo

SUMMARY:
Cell-free hemoglobin can be measured in the plasma of patients with sickle cell anemia, hemodialysis, after red blood cell transfusion, and in patients with sepsis. Cell-free hemoglobin in these patient population has been associated with poor outcomes, including an association with an increased risk of death. Acetaminophen may have a protective effect in these patient populations by inhibiting hemoprotein-mediated lipid peroxidation. The purpose of the present trial is to study the effect of acetaminophen on lipid peroxidation in adults with severe sepsis and detectable cell-free hemoglobin.

The primary hypothesis is that systemic markers of oxidative stress and lipid peroxidation, as measured by F2-isoprostanes, will be significantly lower in patients with severe sepsis and detectable cell-free hemoglobin who receive acetaminophen compared to placebo. The secondary hypothesis is that patients with severe sepsis and detectable cell-free hemoglobin treated with acetaminophen will have better clinical outcomes, including decreased incidence of acute kidney injury and lower rates of hospital mortality, compared to those who receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and Female >=18 years old
* Admitted to an Intensive Care Unit
* Severe Sepsis
* Detectable plasma cell-free hemoglobin

Exclusion Criteria:

* patients who received acetaminophen in the past 48 hours prior to enrollment
* intolerance or allergy to acetaminophen
* measured AST/ALT >400 U/L in the 24 hours prior to enrollment
* chronic liver disease defined by a Child-Pugh score >4
* cannot swallow or have no enteral feeding access
* patients with no detectable cell-free hemoglobin
* patients transitioned to palliative care
* pregnant patients or women of childbearing potential without a documented pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Patients will receive acetaminophen at the dose of 1 gram by mouth or by enteral feeding tube every six hours for a total of 72 hours.
  Acetaminophen
- Placebo: Patients will receive placebo by mouth or by enteral feeding tube every six hours for 72 hours.
  placebo
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 21 | 23
Completed | 18 | 22
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [41 to 64] | 58.5 [47.5 to 63.5] | 55.5 [44 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: F2-isoprostanes After 72 Hours of Acetaminophen or Placebo
Description: F2-isoprostanes are a marker of oxidative stress, specifically lipid peroxidation.
Time Frame: 72 hours after randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 18 | 22
pg/mL | 33.4 [24.97 to 43.47] | 40.15 [29.67 to 61.8]
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.353, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: In-hospital Mortality
Description: percent of patients who died in the hospital
Time Frame: Patients will be followed through the end of their hospital stay, an average of 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 18 | 22
Participants | 1 | 4

3. Secondary Outcome: Serum Creatinine After 72 Hours of Treatment With Acetaminophen or Placebo
Description: serum creatinine measurements at 72 hours
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 18 | 22
mg/dL | 1.04 [.61 to 1.44] | 1.36 [.83 to 2.02]

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, an average of 4 weeks
Arm/Group | Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen (N=21) | Placebo (N=23)
AST or ALT >400 U/L (Hepatobiliary disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No